CLINICAL TRIAL: NCT01480895
Title: Identification of Risk Factors for DM Type 2 in Women Post GDM Diagnosis and Its Prevention by Changing Life Style
Brief Title: Prevention of Diabetes Mellitus Type 2 in Women Post Gestational Diabetes Mellitus Diagnosis
Acronym: GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Naomi Meyerstein, Dr Naomi Meyerstein M D, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOR452307CTL
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Diabetes Mellitus Type 2; Gestational Diabetes Mellitus; Glucose Intolerance; Physical exercise; Nutritional Habits; Dyslipidemia
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Glucose Intolerance; Motor Activity; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post GDM follow-up group. (No Intervention)
  Interventions: Behavioral: Lifestyle instruction for Jews and Bedouin GDM women.
- lifestyle intervention group. (Experimental): The women in this group had participated in lifestyle intervention by diet instructions and physical exercise program.
  Interventions: Behavioral: Lifestyle instruction for Jews and Bedouin GDM women.

INTERVENTIONS:
Behavioral: Lifestyle instruction for Jews and Bedouin GDM women. — Every several months the women had instructions and checkups.
  Other Names: Jew and Bedouin women with recent GDM in the Negev area.

SUMMARY:
Diabetes Mellitus (DM) is a chronic metabolic disorder with increasing incidence and long term complications. Its incidence differs in various ethnic populations.Gestational DM (GDM) is diagnosed when impaired glucose tolerance (IGT) is first detected during pregnancy. GDM incidence in Jewish and Bedouin women has been rising in recent years. It has been reported in many studies that women who had been diagnosed with GDM are more prone to GDM in their next pregnancies and to DM Type 2.

Appropriate changes in everyday diet and physical exercise may reduce the chances for future GDM and type 2 DM.

The investigators aim was to determine GDM frequency in the Negev area in Jewish and Bedouin populations and to construct a plan for follow up and reduce future problems by changing their life style.

DETAILED DESCRIPTION:
Diabetes Mellitus is a very common chronic metabolic disorder,currently an epidemic with correlation to obesity. DM frequency differs as a function of population characteristics factors. In Israel it is more prevalent in Jews than in Bedouins. However, lately, there has been a rise in DM frequency in the Bedouin population. This rise is probably due to the change in life style from the traditional way of life towards a western one, characterized by change in food habits and decrease in physical activity. This combination may lead to increased body mass index (BMI)and to DM.

Many studies report higher incidence of DM type 2 following Gestational Diabetes Mellitus (GDM). GDM is defined as glucose intolerance which is detected during pregnancy in healthy women. Its frequency varies between 1 to 14% in pregnant women in different populations. Although usually glucose intolerance disappears after delivery,many of these women may develop future GMD or DM type 2. This can be delayed or even prevented by appropriate diet and increased physical activity.

The aim of our study was:

1. To determine GDM frequency in Jewish and Bedouin populations in the Negev area in southern Israel.
2. To approach Jewish and Bedouin GDM women before discharge from the hospital and invite them to join the study and divide them into intervention group and control respectively.
3. To study whether intervention in life style leads to similar results in both populations.
4. To propose a model for predicting persistent lifestyle change intervention.

The study included 180 women diagnosed with GDM ,133 Jewish and 47 Bedouin women.The women were divided in two groups, an intervention group (77 Jewish and 26 Bedouin) and control ones (56 Jewish and 21 Bedouin women). At their first visit, 3 months after delivery all women filled forms about demographic data, nutrition and physical habits. All of them, including the control group were given full information about GDM and increased risk for DM.

All the women signed their informed consent forms for participation in the study. The intervention group had several group meetings every several months. Metabolic parameters were determined, including plasma insulin ,glucose and lipids levels.Height, weight, BMI, blood pressure and abdominal circumference were measured too. The same parameters were determined one and two years post partum. The intervention group had several group meetings every several months with a dietician and a physical exercise instructor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gestational diabetes.

Exclusion Criteria:

* Diabetes Mellitus

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in HOMA ratios (Homeostasis Model Assessments of Insulin Resistance). | Determination of HOMA after one year.
  The metabolic parameters included glucose and insulin levels, to enable calculations of HOMA IR. (Homeostasis Model Assessment of Insulin Resistance).
Change in HOMA. | Detrmination of HOMA after two years.
  HOMA calculations post partum.

SECONDARY OUTCOMES:
Determinations of blood lipids . | Post partum lipids levels after one year.
  Determinations of total lipids , total cholesterol , HDL, LDL and triglycerides levels.
Change in lipids levels after two years post partum. | 2 years after delivery.
  Determinations of total cholesterol, HDL,LDL,and triglycerides after one year.
Post partum BMI changes. | one year after delivery.
  BMI assessments after one year.
BMI changes after delivery. | Two years after delivery.
  BMI assessments after delivery.